CLINICAL TRIAL: NCT02134795
Title: A Pilot Study of a Non-Invasive Neuromodulation Device for Treatment of Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study aimed to enroll 10 patients but only enrolled 6 total. Instead of keeping the study open, it was terminated early with incomplete results.
Sponsor: Scion NeuroStim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00053320
Record Dates: First submitted 2014-05-06; First posted 2014-05-09 (Estimated); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caloric Vestibular Stimulation (CVS) (Experimental): Mild to moderate Parkinson's disease subjects will up to 3 sessions of 19 minutes each with the TNM Device during as many as 2 study visits: 2 sessions separated by 1 hour during the 1st study visit and 1 CVS session during a 2nd study visit.
  Interventions: Device: TNM Device

INTERVENTIONS:
Device: TNM Device — The noninvasive device is worn like a music headset and the patient lies back on a wedge pillow while the device is active. Each session lasts under 20 minutes.

SUMMARY:
This is a single-center, open label study evaluating the acute effect of caloric vestibular stimulation on UPDRS motor scores in Parkinson's Disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient should have a UPDRS motor score of 14 (off medication) or higher (mild to moderate)
* Patient should have a Hoehn & Yahr staging of 1 to 3 (mild to moderate)
* Patient must be an adult (18 years of age or older)

Exclusion Criteria:

* Women who are pregnant or nursing
* have a history of significant cardiovascular disease (no pacemakers)
* have a history of unstable mood disorder or unstable anxiety disorder or psychosis
* use a hearing aid
* have a cochlear implant
* have been diagnosed with neurological disease other than Parkinson's disease. No atypical parkinsonism.
* have a diagnosed vestibular dysfunction
* abuse alcohol or other drugs
* have had eye surgery within the previous three months or ear surgery within the previous six months
* have active ear infections or a perforated tympanic membrane
* have participated in another clinical trial within the last 30 days or are currently enrolled in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Caloric Vestibular Stimulation (CVS)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Caloric Vestibular Stimulation (CVS): ThermoNeuroModulation (TNM) device with a standardized active CVS waveform will be used for all patients. The device will be used twice for ~19 minutes each time. There will be a gap of roughly 1 hour between the two device applications.
  The device is worn like a music headset and the patient lies on a wedge pillow while the device is active. Each session lasts under 20 minutes.
Arm/Group | Caloric Vestibular Stimulation (CVS)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Unknown | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Motor UPDRS Score (Unified Parkinson's Disease Rating Scale)
Description: A motor score prior to use of the device will be established (time zero), the motor test will be repeated after the first use of the device (times 25, 50, and 75 minutes), and then after a second use of the device (times 100, 130, 160 and 220). Any changes in motor scores at the various time points will be noted. A videotape of the motor UPDRS examination will be obtained at baseline and during the final test.
Time Frame: Changes in motor score at 25, 50, 75, 100, 130, 160 and 220 minutes relative to baseline
Population: The study was halted early before any of the participants could complete this endpoint. Therefore, there is no outcome data to analyze.
Arm/Group | Caloric Vestibular Stimulation (CVS)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Caloric Vestibular Stimulation (CVS)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
The study did not achieve full enrollment and was, therefore, halted. This occurred before participants were able to complete outcomes measures, and, therefore, prevented outcome analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No